CLINICAL TRIAL: NCT07397377
Title: Enhancing rTMS Effects Through a State-Dependent Approach - An Intervention for Bradykinesia in Parkinson's Disease
Brief Title: prTMS as an Intervention for Bradykinesia in Parkinson's Disease
Acronym: ADAPT-BK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Research Centre for Magnetic Resonance (Other)
Responsible Party: Principal Investigator, Hartwig R. Siebner, Head of Research, Prof., DMSc, Danish Research Centre for Magnetic Resonance
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2500445
Record Dates: First submitted 2026-01-21; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Bradykinesia; Parkinson Disease
Keywords: Bradykinesia; Basal Ganglia Diseases; Parkinson's Disease; Central Nervous System Diseases; Movement Disorders; Synucleinopathies; Neurodegenerative Diseases; SMA; TMS
MeSH Terms: conditions — Hypokinesia; Parkinson Disease; Basal Ganglia Diseases; Central Nervous System Diseases; Movement Disorders; Synucleinopathies; Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: The study has a double-blinded crossover design . The research participant will, in three separate stimulation sessions, receive either active patterned repetitive transcranial magnetic stimulation (prTMS) before a movement, active prTMS between movements or sham prTMS before a movement. The sessions order will be randomized between research participants. The research participants will be blinded to which treatment they receive at any session.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will receive sham patterned repetitive transcranial magnetic stimulation (prTMS) by flipping the coil upside down. This will still provide similar sensory experience as an active stimulation that the patients will not distinguish between. Bradykinesia assessment is filmed during the visit and an experienced rater is unaware of a treatment condition of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active patterned repetitive transcranial magnetic stimulation (prTMS) before a movement (Active Comparator): Real stimulation with four pulses at the frequency of 200 Hertz (Hz) repeating a 0.2Hz will be delivered on the supplementary motor area (SMA) using the active side of the coil for 30 min. Every burst will be given 100 milliseconds (ms) before a movement.
  Interventions: Device: Active patterned repetitive transcranial magnetic stimulation (prTMS)
- Active patterned repetitive transcranial magnetic stimulation (prTMS) between a movement (Experimental): Real stimulation with four pulses at the frequency of 200 hertz (Hz) repeating a 0.2Hz will be delivered on the supplementary motor area (SMA) using the active side of the coil for 30 min. Every burst will be given between movements.
  Interventions: Device: Active patterned repetitive transcranial magnetic stimulation (prTMS)
- Sham patterned repetitive transcranial magnetic stimulation (prTMS) before a movement (Sham Comparator): Sham stimulation with four pulses at the frequency of 200 hertz (Hz) repeating a 0.2Hz will be delivered on the supplementary motor area (SMA) using the non-active side of the coil for 30 min. Every burst will be 100 milliseconds (ms) before a movement.
  Interventions: Device: Sham patterned repetitive transcranial magnetic stimulation (prTMS)

INTERVENTIONS:
Device: Active patterned repetitive transcranial magnetic stimulation (prTMS) — Transcranial magnetic stimulation (TMS) using Axilum Robotics TMS-Cobot using active side of MagVenture Cool-B65 coil
  Arms: Active patterned repetitive transcranial magnetic stimulation (prTMS) before a movement; Active patterned repetitive transcranial magnetic stimulation (prTMS) between a movement
Device: Sham patterned repetitive transcranial magnetic stimulation (prTMS) — Sham transcranial magnetic stimulation (TMS) using Axilum Robotics TMS-Cobot, flipping the active side of the MagVenture Cool-B65 coil.
  Arms: Sham patterned repetitive transcranial magnetic stimulation (prTMS) before a movement

SUMMARY:
This study investigates the use of patterned repetitive transcranial magnetic stimulation (prTMS) as an intervention for bradykinesia in Parkinson's Disease (PD). More specifically, the study aims to determine whether prTMS over the supplementary motor area (SMA) can reduce severity of bradykinesia in PD patients. This approach may open for more targeted and effective treatment of bradykinesia in PD.

DETAILED DESCRIPTION:
Bradykinesia is one of the core symptoms of Parkinson's Disease (PD) and has multiple facets. Movements become slower and decrease in amplitude. Speed and amplitude of movements decline gradually during repetitive movements, referred to as sequence effect. Spontaneous movements are also reduced, and movement initiation is impaired. These symptoms arise from dysfunction within the brain's motor network, particularly involving the basal ganglia-thalamo-cortical loop. The consequences of bradykinesia are far-reaching, severely affecting the patient's daily life and well-being.

Bradykinesia is primarily treated successfully with pharmacologically dopamine precursor levodopa and/or dopamine agonists. However, not all facets of bradykinesia response to dopamine such as the sequence effect and in addition as disease progresses adverse side effects emerge from medication such as dyskinesia which is involuntary choreiform or dystonic movements. These adverse effects require advanced therapies such as invasive treatment with deep brain stimulation (DBS). However, DBS is highly invasive, expensive, and may come with serious side effects.

Transcranial magnetic stimulation (TMS) has emerged as a promising non-invasive and cost-effective intervention for alleviating bradykinesia. In particular, patterned repetitive TMS (prTMS) over several brain regions including the supplementary motor area (SMA) has shown potential in modulating dysfunctional neural circuits and improving motor symptoms in patients with PD. Recent evidence suggests that the efficacy of prTMS may be enhanced by aligning stimulation with specific brain states, as the brain is most responsive to plasticity-inducing protocols right before a movement.

The current study aims to develop and validate a novel burst-based prTMS protocol called quadri-pulse stimulation (QPS), which consist of high-frequency burst with four pulses in each burst. An excitatory 200 hertz (Hz) QPS protocol has already shown to induce long-lasting plasticity changes and by incorporating the state of the brain the study aim to further enhance the effect of this QPS protocol.

Through a cross-over study design the study will apply active QPS right before a movement, active QPS between movement and sham condition before a movement in patients with PD to determine which produces a meaningful reduction in bradykinesia severity measured by Movement Disorder Society Unified Parkinson's Disease Rating Scale part III (MDS-UPDRS-III) and Modified Bradykinesia Rating Scale (MBRS).

ELIGIBILITY:
Inclusion Criteria:

Above 18 years of age. Clinically established or probable Parkinson's Disease (PD), according to the Movement Disorder Society.

Clinical Diagnostic Criteria for PD. Stable antiparkinsonian medicine for at least four weeks. Signed informed consent.

Exclusion Criteria:

Psychiatric disorders. Current use of antipsychotic medication, Donepezil, or GABAergic agents (e.g., pregabalin, gabapentin).

Frequent benzodiazepine or opioid use defined as more than once per week on a regular basis.

History of neurological disease other than PD. Past or present mental illness. History of epilepsy/conditions associated with increased risk of seizure induction through transcranial magnetic stimulation (TMS).

Close relatives suffering from epilepsy/conditions associated with increased risk of seizures.

Contraindications for magnetic resonance imaging (MRI) Contraindications for TMS Female participants of childbearing age must not be pregnant and must use contraception during the trial.

Refuse to be informed about new health-related information and accidental health-related findings that might appear through participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part III (3.4-3.8) (MDS-UPDRS-III) | Immediately before and after each session of patterned repetitive transcranial magnetic stimulation (prTMS)
  Measure the changes of scores of United Parkinson's Disease Rating Scale Part III in active stimulation compared to sham stimulation. More specifically the bradykinesia scores in 3.4 to 3.8. The total scores range from 0 (good health) to 132 (poor health).
Modified Bradykinesia Rating Scale (MBRS) | Immediately before and after each session of patterned repetitive transcranial magnetic stimulation (prTMS)
  Measure the changes of scores of MBRS in active stimulation compared to sham stimulation. A score from 0 (normale) to 4 (barely perform the excercise) will be given for speed, amplitude and rhythmed in differnet task relating the bradykinesia,

SECONDARY OUTCOMES:
Transcranial evoked potentials (TEPs) | Immediately before and after each session of patterned repetitive transcranial magnetic stimulation (prTMS)
  Change in cortical excitability pre-post stimulation over the SMA
Change from pre- to post patterned repetitive transcranial stimulation (prTMS) in resting-state EEG spectral power in predefined frequency bands | Immediately before and after each session of patterned repetitive transcranial magnetic stimulation (prTMS)
  Spectral power will be quantified in a priori defined frequency bands (e.g., delta, theta, alpha, beta).
Hand Grip Test Battery | Immediately before and after each session of patterned repetitive transcranial magnetic stimulation (prTMS)
  By using grip force devices we will measure:
  * Single grip force both cued and non-cued to test rate of force development and yank
  * Repetitive grip to test sequence effect and fatiguability
Motor Evoked Potentials (MEPs) | Immediately before and after each session of patterned repetitive transcranial magnetic stimulation (prTMS)
  Change in cortical excitability pre-post stimulation measured bilateral from the first dorsal interosseous and tibialis anterior

OTHER OUTCOMES:
Transcranial Magnetic Stimulation Adverse Events and Associated Sensations Questionnaire (TMSens_Q) | Immediately after the patterned repetitive transcranial magnetic stimulation (prTMS) intervention
  Questionnaire for assessing any side effects and sensations associated with TMS stimulation, including the assessment of masking (sham or active treatment) of participants. Each item is rated on a 5-point Likert scale from 0 (no sensation) to 4 (severe sensation), with higher scores indicating worse outcomes.
Non-Motor Symptoms Scale for Parkinson's Disease (NMSS) | Baseline, 4-8 weeks after inclusion
  The Non-Motor Symptoms Scale (NMSS) is a 30-item rater-based scale to assess a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The scores on the NMSS range from 0 to 360, with higher scores implying a higher severity and frequency of nonmotor symptoms.
CANTAB battery | Baseline, 4-8 weeks after inclusion
  Measures of response inhibition, spatial planning and working memory and reaction time
The Parkinson's Disease Questionnaire (PDQ-39) | Baseline, 4-8 weeks after inclusion
  39 item self-administered questionnaire that assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better quality of life.
The World Health Organization Quality of Life (WHOQOL) | Baseline, 4-8 weeks after inclusion
  General quality of life assessment as a part of patient reported outcome assessment. The possible score ranges in each case from 0 to 100 points. Higher scores indicate better quality of life.
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Baseline, 4-8 weeks after inclusion
  Is a clinical scale used to follow the progression of a patient's Parkinson's disease. The total scores range from 0 (good health) to 132 (poor health).

CONTACTS AND LOCATIONS:
Locations (1):
- DRCMR, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Sharing of anonymized data
Time Frame: After study completion
Access Criteria: Anonymized data, reasonable request